CLINICAL TRIAL: NCT05798065
Title: Inpatient Endoscopy Procedure Planning Delays and Impact on Length of Stay and 30-day Readmission
Acronym: Impatience
Status: Not yet recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-16151
Record Dates: First submitted 2023-01-08; First posted 2023-04-04 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Inpatient Endoscopy Delay; Readmission; Prolonged Hospital Stay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Inpatient gastrointestinal endoscopy — all inpatient endoscopy procedures (gastroscopy, colonoscopy, ERCP, sigmoidoscopy) during 2016-2022.

SUMMARY:
Single center retrospective cohort study of all inpatient endoscopy procedures to asses factors associated with inpatient endoscopy delays and impact on length of stay and 30-day readmission

DETAILED DESCRIPTION:
Background: Delays in inpatient endoscopy planning negatively influence the quality and accessibility of care. This may result in higher healthcare costs, negative health outcomes, and unnecessary readmissions and use of hospital beds. Additionally, prolonged hospital stay is associated with poorer health outcomes and risk of nosocomial infections, amongst others.

Objective: To asses factors associated with inpatient endoscopy delays and impact on length of stay and 30-day readmission

Study design: Single center retrospective cohort study of all inpatient endoscopy procedures (gastroscopy, colonoscopy, ERCP, sigmoidoscopy) during 2016-2022. Data will be identified and extracted using CTCue. Only pseudonymized data will be used. Inpatient endoscopy delay will be defined as the number of days between the planned date versus the actual date. Multivariable logistic regression models will be performed to assess factors associated with inpatient endoscopy delay.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years)
* Clinical admission in any hospital department of at least two days during 1 January 2016 and 1 December 2022
* Endoscopic procedure during clinical admission, including gastroscopy, endoscopic retrograde cholangiopancreatography (ERCP), endoscopic ultrasound (EUS), flexible sigmoidoscopy, colonoscopy

Exclusion Criteria:

* Elective admission
* Procedure only for insertion of nasogastric or nasojejunal (feeding) tube without any other diagnostic or therapeutic aims

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult inpatients from all hospital departments undergoing endoscopy procedures. Patients will be selected via CTCue, with an admission based query that selects all adult patients with an admission of at least two days between 1-1-2014 and 1-12-2022 AND an endoscopic care activity.
Sampling Method: Non-Probability Sample
Enrollment: 3700 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of inpatient endoscopy delays (IED) | at endoscopic procedure
  IED will be defined as the number of days between the planned date versus the actual date.
Difference in type of endoscopic procedure between patients with and without IED | at endoscopic procedure
  Type of endoscopic procedure: gastroscopy/colonoscopy/endoscopic retrograde cholangio-pancreaticography (ERCP)
Difference in type of sedation between patients with and without IED | at endoscopic procedure
  Type of sedation during endoscopic procedure: No sedation/conscious sedation/general anesthesia

SECONDARY OUTCOMES:
Median length of hospital stay | through study cohort period from 1 january 2016 until 31 december 2022
  length of hospital admission in days
rate of 30-day readmissions | up to 30 days
  percentage of readmissions within 30 days after initial discharge
Odds ratio of presence of inpatient endoscopy delays for risk of prolonged length of hospital stay and 30-day readmissions | from admission till 30 days after discharge
  multivariable logistic regression modelling to assess factors associated with both outcomes and the impact of inpatient endoscopy delay
Odds ratio of presence of inpatient endoscopy delays for risk of 30-day readmissions | from admission till 30 days after discharge
  multivariable logistic regression modelling to assess factors associated with both outcomes and the impact of inpatient endoscopy delay

CONTACTS AND LOCATIONS:
Overall Officials: Peter Siersema, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon reasonable request
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 15 years after publication date
Access Criteria: supporting information will be shared upon reasonable request